CLINICAL TRIAL: NCT05094323
Title: Analgesic Efficacy of Ultrasound-Guided Deep Serratus Anterior Plane Block, Local Wound Infiltration, and Thoracic Paravertebral Block After Uniportal Video-Assisted Thoracic Surgery: A Randomized Trial
Brief Title: Analgesia After Video-Assisted Thoracic Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Seham Mohamed Moeen Ibrahim, Assistant professor of Anesthesia and Intensive Care, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 10 2021
Record Dates: First submitted 2021-10-14; First posted 2021-10-26 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Active Comparator): Patients will receive ultrasound-guided deep serratus anterior plane block.
  Interventions: Drug: Ultrasound-guided deep serratus anterior plane block with isobaric bupivacaine
- Group II (Active Comparator): Patients will receive local wound infiltration (LWI).
  Interventions: Drug: Local wound infiltration with isobaric bupivacaine
- Group III (Placebo Comparator): Patients will receive ultrasound-guided thoracic paravertebral block.
  Interventions: Drug: Ultrasound-guided thoracic paravertebral block with isobaric bupivacaine

INTERVENTIONS:
Drug: Ultrasound-guided deep serratus anterior plane block with isobaric bupivacaine — Patients will receive ultrasound-guided deep serratus anterior plane block with isobaric bupivacaine.
  Arms: Group I
Drug: Local wound infiltration with isobaric bupivacaine — Patients will receive local wound infiltration with isobaric bupivacaine.
  Arms: Group II
Drug: Ultrasound-guided thoracic paravertebral block with isobaric bupivacaine — Patients will receive ultrasound-guided thoracic paravertebral block with isobaric bupivacaine.
  Arms: Group III

SUMMARY:
Although less invasive, postoperative analgesia remains challenging in patients undergoing uniportal video-assisted thoracic surgery (VATS).

DETAILED DESCRIPTION:
Although less invasive, postoperative analgesia remains challenging in patients undergoing uniportal video-assisted thoracic surgery (VATS).

Adequate postoperative pain relief is imperative to hasten functional recovery, accelerate discharge from the hospital, and reduce chronic postsurgical pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for uniportal VATS under general anesthesia, ASA status I-III, aged from 18 to 70 years old of both sex.

Exclusion Criteria:

* Contraindications to regional block
* Pregnancy
* Body mass index (BMI) > 30 Kg/m2
* Psychiatric diseases
* Severe renal, liver, or cardiac dysfunction

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2022-02-18 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Time to first analgesic requirement | 24 hours after surgery
  Assessed in minutes

SECONDARY OUTCOMES:
Postoperative pain intensity | 24 hours after surgery
  Assessed by the numerical rating pain scale, an 11-point scale graded from 0 to 10 (0 = no pain, 10 = the worst imaginable pain)

CONTACTS AND LOCATIONS:
Overall Officials: Seham M Moeen, MD, Principal Investigator — Assiut University
Locations (1):
- Seham M. Moeen, Asyut, Egypt